CLINICAL TRIAL: NCT07388147
Title: Structural Measures for Multiple Myeloma Patients to Improve Rehabilitation by Exercise Therapy
Brief Title: Exercise Therapy for Multiple Myeloma Patients
Acronym: SAPPHIRE-MM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Ulrike Dapunt, Prof. Dr. med., University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S-561/2025
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma Bone Lesions
Keywords: Implementation of structural measures; Rehabilitation; Exercise therapy; Multiple Myeloma; Bone lesions
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthopedic consultation and exercise to evaluate structural measures and improve rehabilitation (Active Comparator)
  Interventions: Other: Orthopedic consultation and rehabilitation by excercise therapy

INTERVENTIONS:
Other: Orthopedic consultation and rehabilitation by excercise therapy — All patients will receive a continuous orthopaedic consultation on bone stability and recommendations for exercise therapy during the different phases of systemic myeloma therapy. Thereby, structural measures to improve rehabilitation in multiple myeloma will be established and evaluated with the intention of integrating them into routine clinical care.

SUMMARY:
Physical exercise is an important supportive therapy for cancer patients, as it improves quality of life in general and might mitigate the side effects of drug treatment. For patients with multiple myeloma in particular, significantly less evidence on the effectiveness of exercise therapy is available due to the fact that this disease is associated with severe bone degradation which might affect bone stability. Advances in oncologic drug treatment have improved overall survival in multiple myeloma significantly. Therefore, there is an increased interest for recommendations on physical activity in this patient group. Due to uncertainties regarding safety and feasibility of exercise therapy in multiple myeloma, both patients and therapists often remain hesitant. Therefore, an orthopaedic outpatient clinic has been established at the Myeloma Center of Heidelberg University Hospital. Here, patients receive consultation on bone stability and individualized physical exercise plans. Based on the expertise gained at the orthopaedic outpatient clinic, the aim of this study is to establish and evaluate structural measures for improved rehabilitation in multiple myeloma and to integrate them into routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed multiple myeloma
* Survival prognosis > 6 months
* ECOG status ≤ 3
* Age ≥18 years
* Patients who state that they want to carry out the training program at least 2 x/week and participate in the planned follow-up visits
* Ability to give informed consent
* Written consent to participate in the study
* Sufficient knowledge of written and spoken German

Exclusion Criteria:

* physical or mental limitation that would prevent participation in the training program or the planned follow-up visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical function | From enrollment to the end of induction therapy after 18 weeks
  Results of the EORTC QLQ-C30 questionnaire ("Physical functioning" scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Heidelberg University Hospital - GMMG Study Group, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
* questionnaire results of each study participant
  * functional assessment of each study participant